CLINICAL TRIAL: NCT04442451
Title: Mechanisms of Fatigability and the Protective Effects of Exercise in People With Diabetes
Brief Title: Mechanisms of Fatigability With Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Illinois at Chicago (Other); Medical College of Wisconsin (Other); University of Wisconsin, Madison (Other); National Institute on Aging (NIA) (NIH); Marquette University (Other)
Responsible Party: Principal Investigator, Sandra Hunter, Francie Kraker Goodridge Collegiate Professor of Kinesiology and Professor of Kinesiology, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00255375; 5R01AG077688-03 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Pre-diabetes; Type 2 Diabetes
Keywords: Diabetes; Pre-diabetes; Fatigability; Blood Flow Restriction Training; Vascular Function; Muscle Fatigue
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Each participant will attend 3 sessions per week for 8 weeks. A training session will start with a 10-minute warm up on a bike ergometer. Each leg will then perform low-load resistance training (~20% of 1-RM) for 4 sets of contractions with 15 contractions per set of contractions with a 30 second rest between each set of contractions while seated in a knee extension weight machine. One leg will be randomized to always perform the training with blood flow restriction (BFR leg) while the contralateral leg performs the exercise training without blood flow occlusion (Control leg).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Exercise (Experimental): Low-load knee extension resistance training (20% of 1-RM) without blood flow restriction. A 10-cm wide inflatable cuff will be placed around the upper portion of the thigh but not inflated.
  Interventions: Other: Control Exercise
- Blood Flow Restriction Exercise (Experimental): Low-load knee extension resistance training (20% of 1-RM) with blood flow restriction using a 10-cm wide inflatable cuff placed around the most proximal part of the exercising thigh. Blood flow will be restricted in the BFR leg at above the limb occlusion pressure of the and this will be determined prior to the exercise while the participant is seated in the knee extensor machine. The cuff pressure during the BFR protocol will be 10 mmHg above limb occlusion pressure.
  Interventions: Other: Blood Flow Restriction Exercise

INTERVENTIONS:
Other: Control Exercise — Each participant will attend 3 sessions per week for 8 weeks. Participants will perform low-load knee extension resistance training (20% of 1-RM) without blood flow restriction on the designated leg for 4 sets of contractions with 15 contractions per set of contractions with a 30 second rest between each set of contractions.
  Arms: Control Exercise
Other: Blood Flow Restriction Exercise — Each participant will attend 3 sessions per week for 8 weeks. Participants will perform low-load knee extension resistance training (20% of 1-RM) with blood flow restriction on the designated leg for 4 sets of contractions with 15 contractions per set of contractions with a 30 second rest between each set of contractions.
  Arms: Blood Flow Restriction Exercise

SUMMARY:
Pre-diabetes (Pre-D) is a precursor to type 2 diabetes (T2D) and characterized by increased exercise fatigability of lower limb muscles, that can impede exercise performance. The cause for the increased fatigability in people with Pre-D is not known. Given the profound vascular disease present in people who have had uncontrolled diabetes for several years, we will determine whether dynamic, fatiguing contractions of the lower limb muscles in people with Pre-D are limited by vascular dysfunction at multiple levels along the vascular tree including the artery, arteriole, and/or capillary. This clinical trial involves a novel exercise training regime involving blood flow restriction to the exercising limb will be used as a probe to further understand the vascular mechanisms for increased fatigability in people with Pre-D and T2D. The long-term goal is to better understand what limits exercise and functional performance in people with diabetes to help develop targeted, more effective exercise programs.

DETAILED DESCRIPTION:
The aim of the clinical trial is to determine the effectiveness of dynamic resistance exercise training coupled with blood flow restriction to improve fatigability and vascular function in people with Pre-D and T2D. People with Pre-D and T2D from Aim 1 will perform 8 weeks of dynamic unilateral resistance exercise training in which one leg is exercised with freely perfused conditions and the other leg with blood flow restriction.

We will assess fatigability, skeletal muscle metabolism, capillary density, and vascular function in people with Pre-D and T2D before and after a novel training intervention that couples dynamic resistance training with blood flow restriction to the exercising limb. This novel intervention has been shown to improve vascular function in young and older adults but has not been investigated in people with Pre-D and T2D. Endothelial function in intact large conduit arteries and arterioles isolated from skeletal muscle biopsies will be measured before and after the training intervention to assess whether the novel training improves vascular function along multiple levels of the vascular tree in people with Pre-D and T2D. Skeletal muscle blood flow through the femoral artery will be quantified with Doppler ultrasonography and skeletal muscle oxygenation will be measured with near infrared spectroscopy (NIRS) during a dynamic fatiguing knee extension exercise. We will closely match participant groups for physical activity levels, age, sex, and body mass index (BMI), because these confounders are not typically controlled for in other human studies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women adults 30 years to 85 years or less
* Pre-diabetes [glycosylated hemoglobin (HbA1c) of 5.7-6.4% and fasting plasma glucose 100-125 mg/dL at the time of initial screening]
* Controls [normoglycemic with a HbA1c level ≤5.6% and fasting blood glucose ≤ 99 mg/dL (5.5 mmol/L)]
* Type 2 Diabetes Mellitus [elevated glycosylated hemoglobin (HbA1c) >6.5% and <10%]

Exclusion Criteria:

* Signs or symptoms of neuropathy
* Medications associated with advanced stages of T2D including insulin
* Poor glycemic control (HbA1c>10%)
* Peripheral edema
* Severe obesity (BMI, >45kg·m-2)
* Untreated hypothyroidism
* Smoking
* Hypertension
* Cardiovascular or musculoskeletal disease that preclude exercise testing
* Hormone replacement drugs or vasoactive medications

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Fatigability - Reduction in Power | One session before and then after 8 weeks of training
  Reduction in limb power and maximal force in response to a dynamic fatiguing contraction.
Strength - 1 Repetition Maximum | One session before and then after 8 weeks of training
  Reduction in limb power and maximal force in response to a dynamic fatiguing contraction
Strength - Maximal Voluntary Contraction (MVC) | One session before and then after 8 weeks of training
  Changes in MVC after 8 weeks resistance training. MVC is the greatest force generated during a brief isometric contraction.
Leg Blood Flow | One session before and then after 8 weeks of training
  Femoral artery mean blood velocity and femoral artery diameter will be measured using Doppler ultrasonography before and immediately after the fatiguing task in each leg.
Skeletal Muscle Oxygenation | One session before and then after 8 weeks of training
  Near-Infrared Spectroscopy recordings will be used to quantify blood flow kinetics of the knee extensor muscle tissue (rectus femoris and vastus lateralis) during the dynamic, fatiguing exercise in each leg.
Vasodilation in Skeletal Muscle Arterioles | One session before and then after 8 weeks of training
  Vessel diameters of arterioles that are extracted and isolated from Skeletal muscle biopsies of the vastus lateralis will be measured in response to vasodilators and constrictors
Muscle Metabolism - Phosphorus Nuclear Magnetic Resonance Spectroscopy (31P-MRS)) | One session before and then after 8 weeks of training
  31P-MRS is used to noninvasively measure muscle metabolism by calculating intracellular ATP, ADP, phosphocreatine (PCr), inorganic phosphate (Pi), and pH in the quadriceps of participants. This measurement is conducted while participants perform fatiguing knee extensor exercise in the magnetic bore.
Capillary density | One session before and after 8 weeks of training
  Immunohistochemical analysis will be performed on muscle biopsy samples to determine the number and density of capillaries for each fiber type.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared